CLINICAL TRIAL: NCT02928952
Title: Effects of a Mindfulness Intervention Delivered Within Diabetes Education on Diabetes-related Outcomes in Military Veterans
Brief Title: Mindful Stress Reduction in Diabetes Self-management Education for Veterans
Acronym: Mind-STRIDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NRI 15-150
Record Dates: First submitted 2016-10-04; First posted 2016-10-10 (Estimated); Results first posted 2021-05-28 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Diabetes Mellitus
Keywords: Mindfulness; Diabetes Distress
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Diabetes Self Management Education (DSME) + Mind-STRIDE (Experimental): Will receive routine diabetes self-management education + the Mind-STRIDE intervention
  Interventions: Behavioral: Mind-STRIDE
- DSME alone (No Intervention): Usual care control

INTERVENTIONS:
Behavioral: Mind-STRIDE — Mindful Stress Reduction in Diabetes Education- mindfulness training with home practice will be introduced as part of diabetes education
  Arms: Diabetes Self Management Education (DSME) + Mind-STRIDE

SUMMARY:
The purpose of this study is to see if adding Mindfulness training to diabetes education reduces feelings of stress and makes it easier to adhere to healthy behaviors that improve diabetes outcomes (such as hemoglobin A1c).

DETAILED DESCRIPTION:
Background: One million Veterans (25%) who receive health care through Veterans Health Administration (VHA) have diabetes and are therefore responsible for daily diabetes self-management (DSM). DSM is essential for glycemic control and prevention of potentially life threatening and disabling complications such as severe hypoglycemia, kidney failure, acute coronary syndrome and stroke. Importantly, 40% of individuals with diabetes suffer from diabetes-related distress (DRD) that interferes with their ability to sustain healthy self-management behaviors, and may be particularly problematic for Veterans who are at higher risk for comorbid negative emotional states such as depression and post-traumatic stress disorder.

Diabetes self-management education (DSME) has traditionally contained little content or skill-building directly related to stress management, leaving this critical component of diabetes self-management largely unaddressed in DSME. In the investigators' pilot work, the investigators have developed a brief stress management intervention known as Mind-STRIDE, which contains mindfulness training and home practice and is easily integrated into existing DSME. While the investigators have previously demonstrated the feasibility, patient acceptability, and initial efficacy of Mind-STRIDE, its effects on diabetes-related psychological and physiological patient outcomes remain unknown. There is, therefore, a critical need to determine the efficacy of this targeted mindfulness intervention for improving DRD, diabetes self-efficacy, DSM behaviors, and metabolic control of Veterans with diabetes in order to offer comprehensive, evidence-based DSME that improves Veteran-centric diabetes outcomes.

Objectives: The objectives of this study are to determine the efficacy of Mind-STRIDE for improving DRD, diabetes self-efficacy, DSM, and metabolic control, and to characterize distinctive Veteran experiences with DRD and Mind-STRIDE.

Methods: To achieve these objectives, the investigators will conduct a randomized controlled trial of 126 Veterans at a large VA medical center in southwest PA. Participants will be assigned to one of two study conditions: an experimental group that receives routine diabetes education plus Mind-STRIDE, or to a usual care group that receives diabetes education alone. DRD, diabetes self-efficacy, and DSM will be assessed using self-report questionnaires. Metabolic control (Hemoglobin A1c) will be assessed using standard laboratory procedures. Data will be collected at baseline, 12-weeks, and 24-weeks, and will be analyzed using mixed-effects models. Telephone interviews will be conducted at 15-weeks post-intervention in a subset of participants from the experimental group, and will be analyzed using modified Grounded Theory methods. Quantitative and qualitative findings will be compared and interpreted using Convergent Parallel Design.

Status: Assessments were completed 4/09/2020.

ELIGIBILITY:
Inclusion Criteria:

* Referral to DSME class at VA Pittsburgh Healthcare System University Drive Campus (VAPHS UD)
* Diagnosis of type 1 or type 2 diabetes
* Hemoglobin A1C >7.0%
* Problem Areas in "Diabetes Scale (PAID) -5" score =/ >3 or "Diabetes Distress Scale -2" =/>2 score indicating the presence of Diabetes-related Distress

Exclusion Criteria:

* Documented cognitive impairment that would interfere with the ability to comprehend the informed consent and actively participate in the study
* Previous attendance of VA DSME class within the past 12 months
* Currently active mindfulness practice

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2020-04-09 (Actual); Study Completion 2020-04-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monica M. DiNardo, PhD ARNP CDE, Principal Investigator — VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA
Locations (1):
- VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
There are currently no plans to share Individual Participant Data (IPD).

REFERENCES:
- [Derived] DiNardo MM, Greco C, Phares AD, Beyer NM, Youk AO, Obrosky DS, Morone NE, Owen JE, Saba SK, Suss SJ, Siminerio L. Effects of an integrated mindfulness intervention for veterans with diabetes distress: a randomized controlled trial. BMJ Open Diabetes Res Care. 2022 Mar;10(2):e002631. doi: 10.1136/bmjdrc-2021-002631. PMID 35346971

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment: 11-1-2016 to 10-31-2019 Diabetes outpatient clinic at VA Pittsburgh Healthcare System, Oakland campus
Pre-assignment Details: One participant was excluded because of concomitant enrollment in a similar study that could have confounded results.
Period: Overall Study
Arm/Group | Diabetes Self Management Education (DSME) + Mind-STRIDE | DSME Alone
Started | 65 | 67
Completed | 55 | 60
Not Completed | 10 | 7
Not completed — Lost to Follow-up | 5 | 5
Not completed — Withdrawal by Subject | 5 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Diabetes Self Management Education (DSME) + Mind-STRIDE | DSME Alone | Total
Number analyzed (Participants) | 65 | 67 | 132
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (10.5) | 60.7 (10.8) | 60.7 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 60 | 61 | 121
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 20 | 23 | 43
  White | 45 | 44 | 89
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 65 | 67 | 132
Living with partner [Count of Participants; unit: Participants] — Married/living with partner vs living alone
  Participants | 26 | 31 | 57
Post-High School Education [Count of Participants; unit: Participants] | 54 | 52 | 106
Employment Status- working full or part time [Count of Participants; unit: Participants] | 18 | 14 | 32
Diabetes Phenotype-type 2 diabetes [Count of Participants; unit: Participants] | 62 | 62 | 124
Charlson Co-Morbidity Index (CMI) [Mean (Standard Deviation); unit: units on a scale] — Comorbidity: 21-item Charlson Comorbidity Index (CCI) predicts one-year mortality based on age range (<40=0;>70=4), and comorbid conditions (e.g. diabetes with/without complications; MI, stroke, solid tumor with/ without metastasis). Each condition is assigned a score of 1 to 6 depending on the magnitude of its associated1-yr mortality risk. Scores are summed and range from a minimum Score of 1 (since all participants had diabetes) to a maximum of 37 for highest risk for age and each condition. Higher scores reflect greater risk, with scores ≥5 representing more severe risk.
  units on a scale | 4.31 (141) | 4.33 (1.79) | 4.32 (1.61)
Insulin use [Count of Participants; unit: Participants] — Diabetes medications: insulin vs. non-insulin use
  Participants | 46 | 47 | 93
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 12.09 (9.67) | 13.81 (11.05) | 12.96 (10.39)

OUTCOME MEASURES:

1. Primary Outcome: Problem Areas in Diabetes Scale (PAID) -(Measures Diabetes Distress)
Description: A 20-item psychometrically validated self-report questionnaire on a 5 point Likert scale (0= not problem; 4= a serious problem). The scores are summed and multiplied by 1.25. Minimum value = 0; Maximum value = 100. Higher scores denote higher levels of diabetes related distress. The cutoff for significant distress is 33; a score of 40 is consistent with diabetes burn-out.
Time Frame: baseline, 12 weeks and 24 weeks
Population: Numbers analyzed differ among rows from the overall number analyzed because of attrition and missed visits.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Diabetes Self Management Education (DSME) + Mind-STRIDE | DSME Alone
Number analyzed (Participants) | 65 | 67
units on a scale
  Baseline | 27.58 (15.41) | 31.24 (16.72)
  12 weeks: number analyzed (Participants) | 51 | 61
  12 weeks | 17.00 (13.10) | 20.83 (13.32)
  24 weeks: number analyzed (Participants) | 55 | 60
  24 weeks | 12.89 (11.30) | 21.15 (13.02)
Statistical Analysis 1: Comparison: Diabetes Self Management Education (DSME) + Mind-STRIDE vs DSME Alone; The statistical analysis was applied to both groups; Test type: Superiority — Assessed group by time differences from week 12 to week 24. Statistical Test of hypothesis. Analyzed as intention to treat in mixed models with imputation as last value moved forward; p = 0.153, Mixed Models Analysis; All models adjusted for Age and Duration of Diabetes
Statistical Analysis 2: Comparison: Diabetes Self Management Education (DSME) + Mind-STRIDE vs DSME Alone; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.026, Mixed Models Analysis; Adjusted for age and duration of diabetes
Statistical Analysis 3: Comparison: Diabetes Self Management Education (DSME) + Mind-STRIDE vs DSME Alone; Within group analysis of intervention effect on Diabetes Distress (Problem Areas in Diabetes, PAID scale) over time stratified by hemoglobin A1c<8.5% and =/>8.5; Test type: Superiority — Analyzed as intention to treat in mixed models with imputation as last value moved forward; p = 0.012, Mixed Models Analysis; Models adjusted for age and duration of diabetes

2. Secondary Outcome: Diabetes Self-efficacy Scale (DSES)
Description: An 8-item psychometrically validated self-report questionnaire on a 10- point Likert Scale (1= Not confident at all; 10 = Totally confident). This scale measures diabetes self efficacy, a critical pathway to improved self-management that refers to an individual's confidence in their ability to perform key diabetes self-management behaviors. Scores are derived as the mean of the 8 questions. Minimum score =1; Maximum Score = 10. Higher scores denote higher diabetes self-efficacy.
Time Frame: baseline, 12 weeks and 24 weeks
Population: Statistical Test of hypothesis. Differing sample sizes are due to attrition and missed research visits. Analyzed as intention to treat in mixed models with imputation as last value moved forward.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Diabetes Self Management Education (DSME) + Mind-STRIDE | DSME Alone
Number analyzed (Participants) | 65 | 67
score on a scale
  Baseline | 6.20 (1.94) | 5.77 (1.95)
  12 weeks: number analyzed (Participants) | 51 | 61
  12 weeks | 6.97 (1.91) | 6.40 (1.80)
  24 weeks: number analyzed (Participants) | 55 | 60
  24 weeks | 7.26 (2.10) | 6.47 (1.92)
Statistical Analysis 1: Comparison: Diabetes Self Management Education (DSME) + Mind-STRIDE vs DSME Alone; Statistical Test of hypothesis. Analyzed as intention to treat in mixed models with imputation as last value moved forward; Test type: Superiority — The statistical analysis was applied to both groups; p = .604, Mixed Models Analysis; All models adjusted for age and duration of diabetes

3. Secondary Outcome: Hemoglobin A1c (A1C)
Description: A blood test that measures the percentage of glycated hemoglobin in red blood cells as a means of estimating the average blood sugar concentrations for the preceding two to three months. Lower percentage denote better blood glucose levels and may range from 4.5% in persons without diabetes t0 >15% in persons with poorly managed hyperglycemia. . An A1C <7% has been associated with prevention of diabetes complications. A1C>9% denotes chronic,severe blood glucose elevation. All tests were performed at VAPHS according to National Glyco-hemoglobin Standardization Program-approved methods.
Time Frame: baseline, 12 weeks and 24 weeks
Population: Number analyzed differs in one or more rows from overall number analyzed due to attrition, missed research assessment, missed visit or failure to go to the lab to have bloodwork done following the research assessment. Three participant in the intervention group and 2 participants in the DSME-alone group did not have A1C done following the 24 week assessment related to closure of the outpatient lab due to COVID-19.
  Analyzed as intention to treat with imputation moving last value forward.
Measure: Mean (Standard Deviation); unit: percentage of glycated Hemoglobin
Arm/Group | Diabetes Self Management Education (DSME) + Mind-STRIDE | DSME Alone
Number analyzed (Participants) | 65 | 67
percentage of glycated Hemoglobin
  Baseline | 8.57 (1.49) | 8.68 (1.63)
  12 weeks: number analyzed (Participants) | 52 | 61
  12 weeks | 7.87 (1.23) | 7.94 (1.22)
  24 weeks: number analyzed (Participants) | 52 | 58
  24 weeks | 7.84 (1.38) | 8.09 (1.51)
Statistical Analysis 1: Comparison: Diabetes Self Management Education (DSME) + Mind-STRIDE vs DSME Alone; The statistical analysis was applied to both groups; Test type: Superiority — Statistical Test of hypothesis. Analyzed as intention to treat in mixed models with imputation as last value moved forward; p = 0.911, Mixed Models Analysis; All models adjusted for Age and Duration of Diabetes

4. Secondary Outcome: Mindfulness Attention and Awareness Scale (MAAS)
Description: A 15-item psychometrically validated questionnaire on a 6-point Likert scale (1=Almost Always and 6= Never) The scale is scored by computing the mean of the 15 items. (Minimum score = 1; maximum score = 6). Higher scores reflect higher levels of dispositional (trait) mindfulness. Average score in the general US population is 4.22. Mindfulness is a mental state achieved by focusing one's awareness on the present moment, while calmly acknowledging and accepting one's feelings, thoughts, and bodily sensations.
Time Frame: baseline, 12 weeks and 24 weeks
Population: Number analyzed differs in one or more rows from overall number analyzed due to attrition and missed or abbreviated visit. One participant had to leave the 24 week visit after completing just 3 of the questionnaires and before completing the other questionnaires. He was then lost to follow-up. He was retained in the Intention-to-Treat analysis since 3 assessments including the primary outcome assessment were completed.
  Analyzed as intention to treat with imputation moving last value forward.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Diabetes Self Management Education (DSME) + Mind-STRIDE | DSME Alone
Number analyzed (Participants) | 65 | 67
score on a scale
  Baseline | 4.37 (0.93) | 4.25 (0.85)
  12 weeks: number analyzed (Participants) | 51 | 61
  12 weeks | 4.49 (0.96) | 4.42 (0.85)
  24 weeks: number analyzed (Participants) | 54 | 59
  24 weeks | 4.52 (1.04) | 4.47 (0.96)
Statistical Analysis 1: Comparison: Diabetes Self Management Education (DSME) + Mind-STRIDE vs DSME Alone; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.940, Mixed Models Analysis; All models were adjusted for age and duration of diabetes

5. Secondary Outcome: Body Weight
Description: Weight in pounds
Time Frame: baseline, 12 weeks and 24 weeks
Population: Number analyzed differs in one or more rows from overall number analyzed due to attrition or missed visit.
  Analyzed as intention to treat with imputation moving last value forward.
Measure: Mean (Standard Deviation); unit: Pounds
Arm/Group | Diabetes Self Management Education (DSME) + Mind-STRIDE | DSME Alone
Number analyzed (Participants) | 65 | 67
Pounds
  Baseline | 227.80 (40.14) | 233.64 (50.15)
  12 weeks: number analyzed (Participants) | 51 | 61
  12 weeks | 229.16 (38.97) | 231.24 (48.29)
  24 weeks: number analyzed (Participants) | 54 | 60
  24 weeks | 229.63 (38.92) | 231.04 (49.53)
Statistical Analysis 1: Comparison: Diabetes Self Management Education (DSME) + Mind-STRIDE vs DSME Alone; The statistical analysis was applied to both groups; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.305, Mixed Models Analysis; All models adjusted for Age and Duration of Diabetes

6. Secondary Outcome: Blood Pressure
Description: Change in mean arterial blood pressure, calculated as blood pressure + 2 (diastolic blood pressure) divided by 3.
Time Frame: baseline, 12 weeks and 24 weeks
Population: Number analyzed differs in one or more rows from overall number analyzed due to attrition, missed visit or shortened visit. Two participants did not have their BP taken at week 24 due to social distancing and COVID-19 precautions.
  Analyzed as intention to treat with imputation moving last value forward.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Diabetes Self Management Education (DSME) + Mind-STRIDE | DSME Alone
Number analyzed (Participants) | 65 | 67
mmHg
  Baseline | 99.46 (12.04) | 100.26 (13.59)
  12 weeks: number analyzed (Participants) | 51 | 61
  12 weeks | 98.51 (13.02) | 95.77 (13.82)
  24 weeks: number analyzed (Participants) | 53 | 60
  24 weeks | 99.61 (13.90) | 96.85 (13.51)
Statistical Analysis 1: Comparison: Diabetes Self Management Education (DSME) + Mind-STRIDE vs DSME Alone; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.228, Mixed Models Analysis; All models adjusted for age and duration of diabetes

7. Secondary Outcome: Patient Health Questionnaire (PHQ8)
Description: The Patient Health Questionnaire (PHQ-8) is a standardized, validated scale that assesses 8 key symptoms of depression experienced over the prior two weeks on a 4-point Likert scale (0=not at all; 3= nearly every day). It is the same as the PHQ-9, without the question regarding suicidal ideation. Score is the sum of the 8 items (Minimum value =0; Maximum= 24). A score of 10 or greater is considered major depression, 20 or more is severe major depression.
Time Frame: baseline, 12 weeks and 24 weeks
Population: Number analyzed differs in one or more rows from overall number analyzed due to attrition, missed visit or missed assessments.One participant had to leave the 24 week visit after completing just 3 of the questionnaires. He was then lost to follow-up. He was retained in the Intention-to-Treat analysis since 3 assessments including the primary outcome assessment (PAID) were completed.
  Analyzed as intention to treat with imputation moving last value forward.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Diabetes Self Management Education (DSME) + Mind-STRIDE | DSME Alone
Number analyzed (Participants) | 65 | 67
score on a scale
  Baseline | 8.22 (5.66) | 9.07 (5.78)
  12 weeks: number analyzed (Participants) | 51 | 61
  12 weeks | 5.98 (5.05) | 6.97 (4.96)
  24 weeks: number analyzed (Participants) | 54 | 60
  24 weeks | 5.61 (5.46) | 7.20 (4.79)
Statistical Analysis 1: Comparison: Diabetes Self Management Education (DSME) + Mind-STRIDE vs DSME Alone; The statistical analysis was applied to both groups; Test type: Superiority — Statistical Test of hypothesis. Differing sample sizes are due to attrition and missed research visits. Analyzed as intention to treat in mixed models with imputation as last value moved forward; p = 0.671, Mixed Models Analysis; All models were adjusted for age and duration of diabetes

8. Secondary Outcome: PTSD Checklist- Civilian Version (PCL-C)
Description: The Abbreviated PCL-C is a validated 6-item civilian version of the PTSD check- list designed for use in general medical settings to assess symptoms of PTSD using a 5-point Likert scale. Scores reflect how much the participant has been bothered by specific PTSD symptoms during the past month. (0= "not at all; 4= "extremely") .Scores are summed. (Minimum value =0; maximum values = 24). Scores >14 are suggestive of PTSD, with higher scores reflecting greater PTSD symptoms.
Time Frame: baseline, 12 weeks and 24 weeks
Population: Number analyzed differs in one or more rows from overall number analyzed due to attrition, missed or incomplete assessments. One participant left the 24- week visit early after completing just 3 of the questionnaires. He was then lost to follow-up. He was retained in the Intention-to-Treat analysis since 3 assessments including that for the primary outcome assessment were completed.
  Analyzed as intention to treat with imputation moving last value forward.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Diabetes Self Management Education (DSME) + Mind-STRIDE | DSME Alone
Number analyzed (Participants) | 65 | 67
score on a scale
  Baseline | 13.22 (5.71) | 13.90 (5.69)
  12 weeks: number analyzed (Participants) | 51 | 61
  12 weeks | 11.63 (4.87) | 12.49 (5.15)
  24 weeks: number analyzed (Participants) | 54 | 60
  24 weeks | 11.09 (5.71) | 12.62 (5.03)
Statistical Analysis 1: Comparison: Diabetes Self Management Education (DSME) + Mind-STRIDE vs DSME Alone; The statistical analysis was applied to both groups; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.571, Mixed Models Analysis; All models were adjusted for age and duration of diabetes

9. Secondary Outcome: Summary of Diabetes Self-Care Activities (SDSCA), General Diet
Description: A 2-item subscale of the psychometrically validated SDSCA that measures the frequency of general dietary behaviors each day over the past 7-days and number of days per week over the past month (0= no days; 7 = 7 days). Scores = mean number of days per week ( Minimum score =0; maximum score = 7) . Higher scores denote healthier dietary behaviors.
Time Frame: baseline, 12 weeks and 24 weeks
Population: Number analyzed differs in one or more rows from overall number analyzed due to attrition or missed visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Diabetes Self Management Education (DSME) + Mind-STRIDE | DSME Alone
Number analyzed (Participants) | 65 | 67
score on a scale
  Baseline | 3.25 (2.07) | 3.51 (1.90)
  12 week: number analyzed (Participants) | 51 | 61
  12 week | 4.60 (1.83) | 4.20 (1.51)
  24 weeks: number analyzed (Participants) | 55 | 60
  24 weeks | 4.93 (1.51) | 3.88 (1.86)
Statistical Analysis 1: Comparison: Diabetes Self Management Education (DSME) + Mind-STRIDE vs DSME Alone; The statistical analysis was applied to both groups; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.003, Mixed Models Analysis; All models adjusted for age and duration of diabetes

10. Secondary Outcome: Summary of Diabetes Self-Care Activities (SDSCA), Specific Diet
Description: A 2-item subscale of the psychometrically validated SDSCA that measures the frequency of eating fruits and vegetables and high fat foods each day over the past 7-days. Minimum maximum values = (0= no days; 7 = 7 days). 1 item is scored as mean number of days (Minimum score =0; maximum score = 7), while the 2nd item is summed and reversed (0= 7days; 7= 0 days). The scores for the two items are summed for the subscale score (Minimum score=0; maximum score =7) Higher scores denote healthier dietary behaviors.
  Each subscale of the SDSCA is scored separately, without a calculated composite score.
Time Frame: baseline, 12 weeks and 24 weeks
Population: Differing sample sizes are due to attrition and missed research visits.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Diabetes Self Management Education (DSME) + Mind-STRIDE | DSME Alone
Number analyzed (Participants) | 65 | 66
score on a scale
  Baseline | 3.28 (1.62) | 2.97 (3.57)
  12 weeks: number analyzed (Participants) | 51 | 61
  12 weeks | 3.71 (1.39) | 3.57 (1.39)
  24 weeks: number analyzed (Participants) | 55 | 60
  24 weeks | 4.01 (1.40) | 3.55 (1.45)
Statistical Analysis 1: Comparison: Diabetes Self Management Education (DSME) + Mind-STRIDE vs DSME Alone; The statistical analysis was applied to both groups; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.632, Mixed Models Analysis; All models adjusted for age and duration of diabetes

11. Secondary Outcome: Summary of Diabetes Self-Care Activities (SDSCA) Space Carbohydrates
Description: One item from the SDSCA that assesses the number of days over the past 7-days in which the participant spaced carbohydrates evenly throughout the day. Minimum score 0; maximum score 7. Higher scores denote healthier dietary behaviors.
Time Frame: baseline, 12 weeks and 24 weeks
Population: Differing sample sizes are due to attrition and missed research visits.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Diabetes Self Management Education (DSME) + Mind-STRIDE | DSME Alone
Number analyzed (Participants) | 65 | 67
score on a scale
  Baseline | 2.91 (2.45) | 2.64 (2.04)
  12 weeks: number analyzed (Participants) | 51 | 61
  12 weeks | 3.76 (1.95) | 3.51 (2.17)
  24 weeks: number analyzed (Participants) | 55 | 60
  24 weeks | 4.42 (1.99) | 3.43 (2.28)
Statistical Analysis 1: Comparison: Diabetes Self Management Education (DSME) + Mind-STRIDE vs DSME Alone; The statistical analysis was applied to both groups; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.219, Mixed Models Analysis; All models were adjusted for age and duration of diabetes

12. Secondary Outcome: Summary of Diabetes Self-Care Activities (SDSCA)- Exercise
Description: A 2-item subscale of the SDSCA that measures the number of days over the past 7-days on which the participant engaged in physical activity . Score = mean score of days over the past 7 days (Min.=1; Max.=7). Higher scores denote healthier exercise behaviors.
  Each SDSCA subscale scored separately.
Time Frame: baseline, 12 weeks, 24 weeks
Population: Differing sample sizes are due to attrition and missed research visits.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Diabetes Self Management Education (DSME) + Mind-STRIDE | DSME Alone
Number analyzed (Participants) | 65 | 67
score on a scale
  Baseline | 2.82 (2.09) | 2.49 (2.06)
  12 weeks: number analyzed (Participants) | 51 | 61
  12 weeks | 3.04 (2.24) | 3.02 (2.33)
  24 weeks: number analyzed (Participants) | 55 | 60
  24 weeks | 3.31 (2.10) | 3.09 (2.31)
Statistical Analysis 1: Comparison: Diabetes Self Management Education (DSME) + Mind-STRIDE vs DSME Alone; The statistical analysis was applied to both groups; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.931, Mixed Models Analysis; All models were adjusted for age and duration of diabetes

13. Secondary Outcome: Summary of Diabetes Self-Care Activities (SDSCA)- - Footcare
Description: A 2-item subscale of the SDSCA that measures the number of days the participant 1) inspected their feet and 2) inspected the inside of their shoes over the past 7-days. Score = mean number of days (Min=0; max=7). Higher scores denote healthier footcare behaviors.
Time Frame: baseline, 12 weeks, 24 weeks
Population: Differing sample sizes are due to attrition and missed research visits.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Diabetes Self Management Education (DSME) + Mind-STRIDE | DSME Alone
Number analyzed (Participants) | 65 | 67
score on a scale
  Baseline | 3.57 (2.30) | 4.04 (2.42)
  12 weeks: number analyzed (Participants) | 51 | 61
  12 weeks | 4.58 (2.18) | 4.81 (2.13)
  24 weeks: number analyzed (Participants) | 55 | 60
  24 weeks | 4.70 (2.25) | 4.85 (2.21)
Statistical Analysis 1: Comparison: Diabetes Self Management Education (DSME) + Mind-STRIDE vs DSME Alone; The statistical analysis was applied to both groups; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.627, Mixed Models Analysis; All models were adjusted for age and duration of diabetes

14. Secondary Outcome: Summary of Diabetes Self-Care Activities (SDSCA)- Blood Glucose Testing
Description: A 2-item subscale of the SDSCA that measures 1) the number of days on which the participant tested their blood glucose over the past 7 days and 2) the number of days on which they tested their blood glucose according to the number of times recommended by their health care provider over the past 7-days. Scores= mean number of days per week. Minimum score is 0 Maximum score is 7.Higher scores denote healthier self-monitoring behaviors.
  Each SDSCA subscale scored separately
Time Frame: baseline, 12 weeks, 24 weeks
Population: Differing sample sizes are due to attrition and missed research visits or skipped questionnaires. One person in each group did not complete the questionnaire at baseline because they were not prescribed blood glucose monitoring by their diabetes care providers.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Diabetes Self Management Education (DSME) + Mind-STRIDE | DSME Alone
Number analyzed (Participants) | 64 | 66
score on a scale
  Baseline | 4.68 (2.71) | 4.94 (2.54)
  12 weeks: number analyzed (Participants) | 51 | 59
  12 weeks | 5.00 (2.50) | 4.92 (2.19)
  24 weeks: number analyzed (Participants) | 54 | 60
  24 weeks | 5.19 (2.33) | 4.56 (2.53)
Statistical Analysis 1: Comparison: Diabetes Self Management Education (DSME) + Mind-STRIDE vs DSME Alone; The statistical analysis was applied to both groups; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.60, Mixed Models Analysis; All models were adjusted for age and duration of diabetes

15. Secondary Outcome: Summary of Diabetes Self-Care Activities (SDSCA)- - Smoking
Description: A 2-item subscale of the SDSCA that measures 1) whether the participant smoked even a puff of a cigarette in the past 7 days (0=no; 1= yes) and 2) if so, the number of cigarettes smoked on an average day. The scores are summed. Minimum score =0, maximum score = >40. Lower scores denote healthier smoking behaviors.
Time Frame: baseline,12 weeks, 24 weeks
Population: Differing sample sizes are due to attrition and missed research visits or incomplete assessment. Two participants in the DSME + Mind-STRIDE intervention group did not complete the Smoking subset of the SDSCA because they do not smoke.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Diabetes Self Management Education (DSME) + Mind-STRIDE | DSME Alone
Number analyzed (Participants) | 63 | 67
score on a scale
  Baseline | 2.82 (5.79) | 2.69 (6.14)
  12 weeks: number analyzed (Participants) | 51 | 61
  12 weeks | 2.13 (5.65) | 3.03 (6.52)
  24 weeks: number analyzed (Participants) | 54 | 58
  24 weeks | 2.12 (6.45) | 2.83 (6.74)
Statistical Analysis 1: Comparison: Diabetes Self Management Education (DSME) + Mind-STRIDE vs DSME Alone; The statistical analysis was applied to both groups; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.461, Mixed Models Analysis; All models were adjusted for age and duration of diabetes

16. Secondary Outcome: Summary of Diabetes Self-Care Activities (SDSCA)- - Medication Adherence
Description: A 2-item subscale of the SDCSA that measures the frequency of 1) taking prescribed insulin and 2)prescribed number of diabetes pills each day over the past 7-days. Scores from the 2 items are summed. Minimum score =0; maximum score = 7). Higher scores denote greater adherence to diabetes medications. Participants entered N/A if they were not prescribed insulin or diabetes pills.
  Each subscale of the SDSCA is scored independently with no calculated composite score.
Time Frame: baseline, 12 weeks, 24 weeks
Population: Differing sample sizes are due to attrition, missed research visits or missing assessment questions. One person in Usual Care Control Group did not take any diabetes medications as reflected in the overall number of participants analyzed in that group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Diabetes Self Management Education (DSME) + Mind-STRIDE | DSME Alone
Number analyzed (Participants) | 65 | 66
score on a scale
  Baseline | 6.49 (1.17) | 6.30 (1.50)
  12 weeks: number analyzed (Participants) | 51 | 61
  12 weeks | 6.28 (1.79) | 6.02 (1.76)
  24 weeks: number analyzed (Participants) | 53 | 57
  24 weeks | 6.45 (1.52) | 6.28 (1.60)
Statistical Analysis 1: Comparison: Diabetes Self Management Education (DSME) + Mind-STRIDE vs DSME Alone; The statistical analysis was applied to both groups; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.906, Mixed Models Analysis; All models were adjusted for age and duration of diabetes

17. Other Pre Specified Outcome: Change in 6-item PROMIS Short Form v1.0 Pain Interference 6 b
Description: A psychometrically validated 7-item instrument on a 5 point Likert scale (1= "not at all"- 5 and "very much") determining the degree to which pain has interfered with aspects of daily living during the past 7 days. It is a general and not disease-specific measure of pain. Scores are summed (Min. value = 6; Max value =35). Total raw scores are then converted into a T-score for each participant. The T-scores rescales the raw score into a standardized score with a mean of 50 and a standard deviation of 10. A score of 50 is the average for the United States general population with a standard deviation of 10.
Time Frame: baseline, 12 weeks and 24 weeks
Population: Number analyzed differs in one or more rows from overall number analyzed due to attrition, missed visits, or skipped assessments. One participant had to leave the 24 week before completing the Pain Interference assessment. He was then lost to follow-up. He was retained in the Intention-to-Treat analysis because he completed 3 of the other assessments including the primary outcome assessment..
  Analyzed as intention to treat with imputation moving last value forward.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Diabetes Self Management Education (DSME) + Mind-STRIDE | DSME Alone
Number analyzed (Participants) | 65 | 67
score on a scale
  Baseline | 56.68 (9.30) | 58.52 (8.64)
  12 weeks: number analyzed (Participants) | 51 | 61
  12 weeks | 54.66 (9.22) | 57.08 (8.78)
  24 weeks: number analyzed (Participants) | 54 | 60
  24 weeks | 53.97 (10.29) | 56.84 (8.31)
Statistical Analysis 1: Comparison: Diabetes Self Management Education (DSME) + Mind-STRIDE vs DSME Alone; The statistical analysis was applied to both groups; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.856, Mixed Models Analysis; All models were adjusted for age and duration of diabetes

18. Other Pre Specified Outcome: Insomnia Severity Index (ISI)
Description: Seven psychometrically tested items on a 4 point Likert scale that measure difficulty falling asleep and staying asleep (0= none; 4=very severe) and satisfaction with current sleep patterns (0=very satisfied; 4=very dissatisfied), Noticeable impairment of quality of life (0= not noticeable; 4= very much noticeable), Worry/distress re: sleep (0=not at all worried; 4=very much worried); Interference of sleep problem to daily functioning (0=not interfering; 4= very much interfering). Scores are summed. Minimum score = 0; maximum score = 20). Higher scores denote greater insomnia severity. Scores over 14 denote insomnia; Scores 8 to 14 denote subthreshold insomnia.
Time Frame: baseline, 12 weeks and 24 weeks
Population: Number analyzed differs in one or more rows from overall number analyzed due to attrition,missed visits or skipped assessments. One participant had to leave the 24 week visit before completing the ISI. He was then lost to follow-up. He was retained in the Intention-to-Treat analysis since he completed 3 of the other assessments including the primary outcome assessment.
  Analyzed as intention to treat with imputation moving last value forward.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Diabetes Self Management Education (DSME) + Mind-STRIDE | DSME Alone
Number analyzed (Participants) | 65 | 67
score on a scale
  Baseline | 11.00 (6.12) | 11.81 (7.51)
  12 weeks | 9.20 (7.15) | 10.34 (6.79)
  24 weeks: number analyzed (Participants) | 54 | 59
  24 weeks | 8.48 (6.48) | 10.14 (7.16)
Statistical Analysis 1: Comparison: Diabetes Self Management Education (DSME) + Mind-STRIDE vs DSME Alone; The statistical analysis was applied to both groups; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.89, Mixed Models Analysis; All models adjusted for age and duration of diabetes

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Diabetes Self Management Education (DSME) + Mind-STRIDE | DSME Alone
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/67
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/67
Other Adverse Events (participants affected / at risk) | 0/65 | 0/67

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-02): https://cdn.clinicaltrials.gov/large-docs/52/NCT02928952/Prot_SAP_000.pdf